CLINICAL TRIAL: NCT07355855
Title: A Multicenter, Multi-cohort, Prospective Phase II Clinical Study on the Efficacy and Safety of All-trans Retinoic Acid Combined With VAC Regimen in the Treatment of Intermediate-to-high-risk Rhabdomyosarcoma
Brief Title: A Clinical Study on the Efficacy and Safety of All-trans Retinoic Acid Combined With VAC Regimen in the Treatment of Intermediate-to-high-risk Rhabdomyosarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Chief Physician, Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMS-ATRA-IIT-01
Record Dates: First submitted 2025-12-30; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATRA+VAC (Experimental)
  Interventions: Drug: ATRA+VAC
- ATRA+VAC+Anlotinib (Experimental)
  Interventions: Drug: ATRA+VAC+Anlotinib

INTERVENTIONS:
Drug: ATRA+VAC — Cohort 1: Intermediate-risk RMS: ATRA+VAC treatment
  The specific medication is:
  Vincristine (V), administered intravenously, at a dose of 1.5 mg/m2 (with a maximum of 2 mg), on days 1, 8, and 15, every three weeks.
  Dactinomycin (A), intravenous infusion, 1.25mg/m2 (maximum not exceeding 2.5mg), D1, q3w.
  Cyclophosphamide (C), intravenous infusion, 1200mg/m2, D1, q3w. All-trans-retinoic acid: provided free of charge by Shandong Liangfu Pharmaceutical Co., Ltd. Capsules, 10mg/capsule, 20mg bid, orally, administered continuously every day, with 21 days constituting one course of treatment. If safety is confirmed, the dosage can be increased to 30mg bid.
  Arms: ATRA+VAC
Drug: ATRA+VAC+Anlotinib — Cohort 2: High risk group RMS+: ATRA+VAC, ATRA+anlotinib maintenance therapy
  The specific medication is:
  Vincristine (V), static push, 1.5 mg/m2 (maximum not exceeding 2mg), D1, 8, 15, q3w.
  Dactinomycin (A), intravenous drip, 1.25mg/m2 (maximum not exceeding 2.5mg), D1, q3w.
  Cyclophosphamide (C), intravenous infusion, 1200mg/m2, D1, q3w. After chemotherapy, Anlotinib, 12mg, d1-d14, po, q3w+ATRA maintenance therapy. Both are maintained for a period of time until disease progression or toxicity is intolerable, or for at least 2 years.
  All trans retinoic acid: provided free of charge by Shandong Liangfu Pharmaceutical Co., Ltd., capsule, 10mg/capsule, 20mg bid orally, administered continuously daily for 21 days as a course of treatment. If safety is ensured, the dosage will be increased to 30mg bid.
  Arms: ATRA+VAC+Anlotinib

SUMMARY:
This study is a prospective, multi-cohort, multi-center clinical trial targeting patients with intermediate-to-high-risk rhabdomyosarcoma who have not previously received systemic anti-tumor treatment. It aims to evaluate the efficacy and safety of all-trans retinoic acid combined with VAC chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 14 years old and ≤ 60 years old;
2. Histologically confirmed medium to high risk rhabdomyosarcoma (excluding pleomorphic rhabdomyosarcoma);
3. The physical fitness status score of the Eastern Cancer Collaboration Group (ECOG) is 0-1;
4. Have not received any anti-tumor drug treatment in the past;
5. Expected survival time ≥ 3 months;
6. Possess sufficient organ and bone marrow function, with laboratory test values meeting the following requirements within 7 days prior to enrollment (no blood components, cell growth factors, albumin, or other corrective treatment drugs are allowed within 14 days prior to obtaining laboratory tests), as follows Blood routine: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin (HGB) ≥ 100 g/L (no transfusion or erythropoietin dependence within 14 days) Liver function: serum total bilirubin ≤ 1.25 times the upper limit of normal (ULN); ALT and AST ≤ 2.5 x ULN (≤ 5x ULN for patients with liver metastases); Serum albumin ≥ 30 g/L; Alkaline phosphatase (ALP) ≤ 5 × ULN.

   Renal function: Serum creatinine (Cr) ≤ 1.25 × ULN, or creatinine clearance rate ≥ 60 mL/min (using the standard Cockcroft Gault formula): Urine routine results show urinary protein<2+; For patients whose baseline urine routine test shows urinary protein ≥ 2+, 24-hour urine collection should be performed with a 24-hour urine protein quantification of<1g.

   Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; If the subject is receiving anticoagulant therapy, as long as the INR is within the intended range of use of the anticoagulant drug.
7. For female subjects of childbearing age, a urine or serum pregnancy test should be conducted 3 days before receiving the first study drug and the result should be negative;
8. Participants and their sexual partners are required to use a medically approved contraceptive measure (such as intrauterine devices, birth control pills, or condoms) during the study treatment period and within 6 months after the end of the study treatment period.

Exclusion Criteria:

1. Previously received anti-tumor treatment other than surgery and radiation therapy for any malignant tumor;
2. Subjects who cannot accept or tolerate this chemotherapy regimen for various reasons;
3. Biopsy confirmed a patient with bone marrow infiltration;
4. Patients who have undergone major surgical procedures unrelated to medium to high risk rhabdomyosarcoma within the 4 weeks prior to enrollment, or who have not fully recovered from such surgical procedures;
5. Serious heart disease or discomfort, including but not limited to the following diseases:

   * Diagnosed history of heart failure or systolic dysfunction (LVEF<50%);
   * High risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate>100bpm, significant ventricular arrhythmias (such as ventricular tachycardia), or higher-level atrioventricular block (i.e. Mobitz II second or third degree atrioventricular block);
   * Angina requiring treatment with anti angina drugs;
   * Clinically significant heart valve disease;
   * ECG shows transmural myocardial infarction;
   * Poor control of hypertension (systolic blood pressure>180mmHg and/or diastolic blood pressure>100mmHg)
6. Individuals with a known history of allergies to the components of this medication regimen;
7. The researcher believes that the patient is not suitable to participate in any other circumstances of this study.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
2-year event-free survival (EFS) rate | up to 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | up to 2 years
Disease control rate (DCR) | up to 2 years
Objective response rate (ORR) | up to 2 years
adverse event | up to 2 years
Quality of life (Functional Assessment of Cancer Therapy - General) | up to 2 years
The correlation between the gene status of PAX3/7-FOXO1 and therapeutic efficacy | up to 2 years
  Subgroup analysis of the effect of PAX3/7-FOXO1 gene expression on the 2-year EFS rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university cancer hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No